CLINICAL TRIAL: NCT03195062
Title: Fructose Extra-splanchnic Metabolism and Its Effects on Systemic Flux of Substrates (FruPP)
Acronym: FruPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, MD, Professor, University of Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-01828
Record Dates: First submitted 2017-03-23; First posted 2017-06-22 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Test Meal
Keywords: Fructose; Obesity; Metabolism; Post-prandial kinetics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test meal (Experimental): The subjects will receive a liquid test meal containing glucose and fructose with 13C fructose.
  Interventions: Other: Test meal

INTERVENTIONS:
Other: Test meal — Liquid test meal (fructose+glucose)

SUMMARY:
In parallel to the dramatic rise in metabolic diseases and diabetes observed over the past fifty years, the generalization of added sugar in processed food led to a marked increase in fructose consumption in almost all countries, and epidemiological studies demonstrated that the consumption of sugar-sweetened beverage (containing at least 50% of fructose) is associated with the development of diabetes, hepatic steatosis, dyslipidemia and obesity.

The objective of the study is to measure the amount of fructose that escape first-pass hepatic extraction after oral ingestion (fructose+glucose), and gain insights into its metabolic fates with the use of tracers.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 40 years
* Body Mass Index of 18.5 to 25 kg/m²
* Sex male of female

Exclusion Criteria:

* Fructose intolerance
* Antidiabetic and hypolipemic drugs
* Alcohol consumption >10g/day
* Severe eating disorders
* Severe psychological problems
* Vegetarian diet or other specific diet
* Consumption of illicit substances
* Pregnancy
* Weight gain or weight loss > 3 kg in the last 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Measurement of the amount of fructose that escape first-pass hepatic extraction after oral ingestion. | The quantity of 13C fructose will be calculated, during the post prandial period, until 240 min.
  Calculation with 13C fructose enrichment in blood samples at T0; 30; 60; 90; 120; 150; 180; 210 and 240 min.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No